CLINICAL TRIAL: NCT01757925
Title: Evaluation of a Commercial Gaming Impact in a Childhood Obesity Intervention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UnitedHealth Group (Industry)
Responsible Party: Principal Investigator, Dr. Deneen Vojta, Dr. Deneen Vojta Vice President of Center for Health Reform and Modernization, UnitedHealth Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JXBX 2012 11-214
Record Dates: First submitted 2012-12-21; First posted 2012-12-31 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-12

CONDITIONS: Childhood Obesity
Keywords: activity; gaming; obesity; Active Gaming; Control
MeSH Terms: conditions — Pediatric Obesity; Motor Activity; Obesity | interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Gaming (Experimental): Participants will receivce a weight management program plus active gaming device
  Interventions: Behavioral: weight managment program; Other: Active Gaming
- Control Group (Active Comparator): Participants will receive a weight management program without active gaming
  Interventions: Behavioral: weight managment program

INTERVENTIONS:
Behavioral: weight managment program — a comprehensive peditric weight management program consisting of 16 weekly group sessions
Other: Active Gaming — partcipants will be given a gaming device and 2 games (1 at baseline and 1 at week 8)
  Other Names: Hands free Kinect gaming device plus 2 games
  Arms: Active Gaming

SUMMARY:
Recently, researchers have been interested in the use of game play, mechanics and psychology for health-related engagement and behavior change. While initial studies have shown some increases in health knowledge and/or behavior through gaming, there remains concern that the vehicle for change is associated with a perceived sedentary behavior (6).

More recently, commercially available gaming devices are able to directly promote physical activity through a new set of "kinetic controllers" added to the gaming experience. UHG plans to evaluate the most recent of these kinetic controller technologies in the context of a second iteration of JOIN (described above) to be implemented among a pilot group of overweight and/or obese children whose BMI percentile is above the 85th.

This study will evaluate the effect of a commercial controller-free Exercise Gaming and Entertainment Experience (EGEE) on physical activity levels in the context of a weight management program in approximately 70 children ages 6 to12. The study will compare the differences in physical activity levels over 16 weeks in two groups of children.

DETAILED DESCRIPTION:
The Center for Health Reform and Modernization at UHG will compare levels of physical activity, assessed by accelerometry, among children randomly assigned to WMA or WM+E groups. Specific aims of this evaluation are:

* Compare the two groups on changes in the daily minutes of physical activity (mild, moderate and vigorous) after sessions 1, 8 and 15, respectively (Sessions are typically one week a part. Due to holiday schedules, there may be a lapse of two weeks between sessions).
* Compare the two groups on changes in the daily minutes of sedentary behavior after sessions 1, 8 and 15, respectively
* Compare the two groups on changes in relative weight (weight, BMI percentile, BMI z-score) at sessions 1, 8, and 16 weeks, respectively
* Compare the two groups on measures of program satisfaction at 1, 8, and 16 weeks, respectively

Participation in the post session one session is required in order to be eligible for the study requirements include:

* A signed consent/ assent from the parent and child.
* The child must be able to participate in physical activity similar to exercise gaming
* The family must have a TV/monitor that supports Microsoft Kinect
* The family must have internet connection in the home

The family's decision to participate in the study does not affect the child's'/ parent's overall ability to fully participate in the JOIN Program. All JOIN program materials will be the same whether or not JOIN participants agree to be in the study. All aspects of the study will be conducted outside of the standard class time. Interested and eligible participants will be scheduled to attend a study visit immediately after their first JOIN class. During that study visit, written informed consent/assent from the parent/child will be obtained.

Once a participant has agreed to enroll and have been consented/assented he/she will be informed of study group to which he/she has been randomly assigned. There are two options: 1) weight management alone or 2) weight management plus exercise gaming and entertainment experience. Randomization will occur at the group level (i.e., all consented/assented children in the Wed at 5 p group). Classes will be randomized in pairs of 2 and based on enrollment.

Treatment JOIN consists of 16 weekly Core in-person group sessions followed by 8 monthly mastery group sessions. While the JOIN Program continues for one year, the study will only occur over the first 16 weeks. YMCA sessions last 75 minutes and include a weight assessment of the child prior to each session. The groups are led by a YMCA facilitator. The topics for the first 16 sessions are listed below.

Child Activity Monitor. At sessions 1, 8, and 15 an actigraph will be distributed to each participating child in group 1 and 2. Each child will wear it for 1 week (7 days) during waking hours, and return it at the next session. An activity monitor provides no feedback to participants and provides an objective measure of physical activity (mild, moderate, vigorous) as well as sedentary behavior through downloaded data. The GT3XE Triaxial Activity Monitor w/Extended Memory® (produced by Actigraph) is a small, omni-directional accelerometer (Actigraph), which has already been approved by the FDA for measuring subject's physical activity, and energy expenditure level. The activity monitor (Actigraph) is a small, 1 inch by 1 inch, device that is worn at the hip level attached to an adjustable belt (also provided by the study). The belt can be worn below or above clothing.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 6 - 12 with Parent or Gaurdian.
* Child must be enroll in JOIN Program,
* Child must have a BMI in the 85th percentile

Exclusion Criteria:

* English Speaking Participants only

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2011-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
MVPA | 16 weeks
  difference between groups in MVPA at week 16 as assess by accelerometry

SECONDARY OUTCOMES:
relative weight | 16 weeks
  difference in % overweight, bmi z-score between groups at week 16
quality of life | 16 weeks
  Differences between groups in pediatric qulaitry of life as assessed by parents and children

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - YMCA Andvore, Andover, Massachusetts
  - YMCA Lawrence, Lawrence, Massachusetts
  - YMCA Merrimack Valley of MAss, Methuen, Massachusetts
  - YMCA Boroughs, Westborough, Massachusetts
  - Barrinton YMCA, Barrington, Rhode Island
  - Newman YMCA, Seakonk, Rhode Island
  - YMCA Kent, Warwick, Rhode Island
  - Jones Elementary, Missouri City, Texas
  - Barabara Jordan Elementary, Richmond, Texas
  - Oyster Creek Elementary, Sugarland, Texas
  - Townwest Elementary, Sugraland, Texas

REFERENCES:
- [Derived] Trost SG, Sundal D, Foster GD, Lent MR, Vojta D. Effects of a pediatric weight management program with and without active video games a randomized trial. JAMA Pediatr. 2014 May;168(5):407-13. doi: 10.1001/jamapediatrics.2013.3436. PMID 24589566